CLINICAL TRIAL: NCT02066948
Title: Effects of Dietary Protein Patterning on wt Loss and Resistance Training-induced Changes in Body Comp, Skeletal Muscle, and Indices of Metabolic Syndrome
Brief Title: Meal Patterning on Weight Loss With Changes to Body Comp, Muscle and Metabolic Health
Acronym: S38
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Collaborators: National Pork Board (Other); American Egg Board (Other); Dairy Research Institute (Other); National Cattlemen's Beef Association, a contractor to the Beef Checkoff (Industry)
Responsible Party: Principal Investigator, Wayne Campbell, Professor, Foods and Nutrition, Purdue University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 1307013804
Record Dates: First submitted 2013-09-12; First posted 2014-02-20 (Estimated); Last update posted 2017-06-01 (Actual); Status verified 2017-01

CONDITIONS: Body Composition, Beneficial; Paresis; Impaired Glucose Tolerance
Keywords: DXA; MRI; Fitness assessment; Meal tolerance test
MeSH Terms: conditions — Glucocorticoid Receptor Deficiency; Paresis; Glucose Intolerance

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Skew meal pattern w/ wt loss&exercise (Active Comparator): Skew meal pattern w/ wt loss&exercise e
  Interventions: Other: wt loss; Other: Meal Pattern; Dietary Supplement: even
- even meal pattern w/ wt loss&exercise (Active Comparator): even meal pattern w/ wt loss&exercise
  Interventions: Other: wt loss; Other: Meal Pattern; Dietary Supplement: skew

INTERVENTIONS:
Other: wt loss — subjects will consume a 750 reduced calorie daily diet based on current ht. wt and age
Other: Meal Pattern — Even or skewed distribution of protein for a 16 week period of wt loss.
Other: meal pattern — skew or even
  Other Names: skew or even
Dietary Supplement: even — even amount of protein distributed between each meal
  Arms: Skew meal pattern w/ wt loss&exercise
Dietary Supplement: skew — a skewed amount of protein is distributed between each meal
  Arms: even meal pattern w/ wt loss&exercise

SUMMARY:
About two-thirds of adults in the United States are overweight or obese with likely adverse health consequences. A Moderate weight loss by dieting and exercise is recommended to improve health. We are interested to know whether eating dietary protein at different times of the day influences changes in body composition, muscle and indices of health. The purpose of this study is to examine the effects of within-day patterning of dietary protein intake (even vs. skewed) on energy-restriction and resistance training-induced changes in body composition, muscle size, appetite, and clinical health (including blood glucose and blood pressure).

DETAILED DESCRIPTION:
About two-thirds of adults in the United States are overweight or obese. Obesity is associated with an increased risk of chronic disease and metabolic syndrome and a reduced physical functioning capacity, all of which contribute to disproportionately high healthcare expenditures and premature mortality. A moderate dietary energy restriction with a higher protein diet has been recommended for weight loss to prevent or improve medical complications associated with obesity as well as improve body composition, including preserving lean body mass. Emerging research indicates that the consumption of multiple high protein meals daily may be superior than only consuming one high-protein meal (typically dinner) to stimulate muscle protein synthesis throughout the day. This concept is based on research showing that the patterning of energy and protein intake influences muscle protein synthesis and whole body composition and protein retention. Very limited research exists regarding the effects of protein intake on skeletal muscle size after weight loss, and currently, no longitudinal studies have evaluated the effectiveness of consuming an even vs. skewed distribution of protein intake across meals on phenotypic changes in skeletal muscle size over the longer-term. Recent studies have also suggested that evenly distributed protein patterning may promote satiety and improve blood glucose response in healthy adult men and women. However, there is a need for controlled, longer-duration trials to investigate the effects of daily protein distribution on appetite, glucose response and metabolic syndrome after weight loss in overweight or obese adults. The goal of the proposed research is to evaluate the effects of within-day patterning of dietary protein intake (even vs. skewed) on energy-restriction and resistance training-induced changes in body composition, skeletal muscle size, appetite, glucose response, and metabolic syndrome parameters.

ELIGIBILITY:
Inclusion Criteria:

* non-smoking;
* weight stable (± 4.5 kg during previous 3 months)
* constant habitual activity patterns within last 3 months
* no acute illness
* not diabetic or have chronic diseases
* blood profile within 10% of clinical normalcy
* subjects not classified as high risk for cardiovascular disease
* no use of medications
* females who are not pregnant or lactating
* ability to travel to testing and exercise training facilities
* not claustrophobic and able to complete the muscle size testing using the magnetic resonance imager

Exclusion Criteria:

* Smoker
* weight changed within 3 months
* a history of disease or high risk of cardiovascular disease
* history of claustrophobic
* pregnant or lactating female

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2014-01; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Body composition | 20 weeks
  Fasting-state body weight and waist and hip circumferences will be measured. Body composition (fat mass, lean body mass, and bone mass) will also be determined using Dual Energy X-ray Absorptiometry (DXA, GE Healthcare LUNAR iDXA™ with EnCORE software version 5.60, Madison, WI).
Body composition | 20 weeks
  Fasting-state body weight and waist and hip circumferences will be measured. Body composition (fat mass, lean body mass, and bone mass) will also be determined using Dual Energy X-ray Absorptiometry

SECONDARY OUTCOMES:
Whole body Imaging | 20 weeks
  A total of 2 magnetic resonance imaging (MRI) images of muscle and 1 MRI of the abdomen will be obtained

OTHER OUTCOMES:
Aerobic Fitness and Muscle Strength Assessment | 20 weeks
  An aerobic fitness will be assessed by submaximal aerobic capacity test and a maximal muscle strength will be examined using a one-repetition maximum test

CONTACTS AND LOCATIONS:
Overall Officials: Wayne W Campbell, Ph.D., Principal Investigator — Purdue University
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

REFERENCES:
- [Derived] Hudson JL, Kim JE, Paddon-Jones D, Campbell WW. Within-day protein distribution does not influence body composition responses during weight loss in resistance-training adults who are overweight. Am J Clin Nutr. 2017 Nov;106(5):1190-1196. doi: 10.3945/ajcn.117.158246. Epub 2017 Sep 13. PMID 28903957